CLINICAL TRIAL: NCT00717886
Title: Upper Extremity Lymphatic Mapping for Breast Cancer Patients: A Pilot Study
Brief Title: Upper Extremity Lymphatic Mapping for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-051
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Axillary Lymph Node Dissection
Keywords: Breast; Lymph Nodes
MeSH Terms: conditions — Breast Neoplasms | interventions — RID; Radioactivity

ARMS (1):
- 1 (Experimental): Patients with documented axillary metastases (Stage II breast cancer) will undergo subdermal injection of technetium sulfur colloid (TSC) into the ipsilateral upper extremity approximately 3 hours before surgery.
  Interventions: Radiation: isosulfan blue dye

INTERVENTIONS:
Radiation: isosulfan blue dye — At the time of surgery, each patient will undergo a subareolar injection of isosulfan blue dye into the ipsilateral breast as routinely performed during a sentinel lymph node mapping for breast cancer. The surgeon will then perform an axillary lymph node dissection in the usual, routine manner. The above differs from standard of care in that patients scheduled for an upfront axillary dissection do not routinely undergo sentinel lymph node mapping- therefore these patients would not normally get any isotope or TSC injections since they already need an ALND. Second, standard sentinel lymph node mapping involves injection of TSC into the affected breast the day prior to surgery or 3 hours before surgery versus injection of TSC into the ipsilateral upper extremity. The protocol specifies "day of" mapping for patient convenience.
  Other Names: Once the specimen is removed from the patient, the axillary nodes will be; dissected from the specimen and categorized: "blue only"; "radioactive only";; "blue and radioactive"; and "neither." The number of axillary nodes which are; "radioactive only" will indicate the nodes which drain the ipsilateral upper; extremity. The "blue and radioactive" nodes will indicate the sentinel lymph; nodes from the breast, which are also nodes that drain the ipstilateral upper; extremity. The prevalence of positive "radioactive only" and /or "blue and; radioactive", "blue only" and nodes with "neither" will be noted.

SUMMARY:
This study is being done to see if lymph nodes that drain the arm also drain the breast. An axillary lymph node dissection removes lymph nodes under the arm. It is done to help prevent cancer cells from spreading to the rest of the body. Usually, about 12 to 15 nodes are removed. They are then examined to see if they have cancer cells. Removing these lymph nodes has some side effects. The most common is lymphedema. This is the build-up of fluid in the arm. This study will tell us if it may be possible in the future to identify lymph nodes that just drain the arm. Leaving those nodes may help to reduce the rate of lymphedema for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Females with Stage II invasive breast cancer and documented axillary metastases by core biopsy, clinical examination, or fine-needle aspiration who are scheduled to undergo an ALND.
* Females > 21 years of age

Exclusion Criteria:

* Prior ipsilateral axillary surgery
* Prior ipsilateral axillary radiation
* Prior ipsilateral breast cancer
* Prior ipsilateral breast radiation
* Allergy to isosulfan blue dye
* History of ipsilateral upper extremity lymphedema
* Prior history of surgical excision of the upper outer quadrant of the ipsilateral breast
* Prior history of neoadjuvant chemotherapy for current breast cancer
* Bulky axillary disease at presentation (N2)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Montgomery, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Upper Extremity Lymphatic Mapping for Breast Cancer Patients: Patients with documented axillary metastases (Stage II breast cancer) will undergo subdermal injection of technetium sulfur colloid (TSC) into the ipsilateral upper extremity approximately 3 hours before surgery.
Period: Overall Study
Arm/Group | Upper Extremity Lymphatic Mapping for Breast Cancer Patients
Started | 13
Completed | 9
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Treatment Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Upper Extremity Lymphatic Mapping for Breast Cancer Patients
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number and Prevalence of Metastases of Blue Nodes in the ALND Specimen (Nodes Draining the Breast).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Upper Extremity Lymphatic Mapping for Breast Cancer Patients
Number analyzed (Participants) | 9
participants | 0

ADVERSE EVENTS:
Arm/Group | Upper Extremity Lymphatic Mapping for Breast Cancer Patients
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes